CLINICAL TRIAL: NCT04267718
Title: Efficacy of the Use of Risk Scores in Reducing Important Clinical Outcomes in Hospitalized Medical Ill Patients: the RICO Cluster-randomized Controlled Trial
Brief Title: Efficacy of the Use of Risk Scores in Reducing Important Clinical Outcomes in Hospitalized Medical Ill Patients
Acronym: RICO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fadoi Foundation, Italy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FADOI.04.2018
Record Dates: First submitted 2019-09-13; First posted 2020-02-13 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Prevention of Venous Thromboembolism

STUDY DESIGN:
Intervention Model Description: The experimental group includes a number of centres that will be randomized to systematically evaluate all eligible patients with the Padua and IMPROVE Bleeding scores within 48 h after hospitalization. The control group includes A number of centres will be randomized to the Control arm of the study, in which patients will be evaluated for their thrombotic and hemorrhagic risk according to clinical judgment only.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with the Padua and IMPROVE Bleeding scores (Experimental): A number of centres will be randomized to systematically evaluate all eligible patients with the Padua and IMPROVE Bleeding scores within 48 h after hospitalization.
  Interventions: Other: Application of Padua and IMPROVE Bleeding scores
- Patients will be evaluated according to clinical judgment only (No Intervention): A number of centres will be randomized to the Control arm of the study, in which patients will be evaluated for their thrombotic and hemorrhagic risk according to clinical judgment only.

INTERVENTIONS:
Other: Application of Padua and IMPROVE Bleeding scores — Eligible patients hospitalized in centres randomized to the Experimental group will be evaluated, within 48 hours from admission to hospital, by means of the Padua predictive score and the IMPROVE Bleeding score.
  Arms: Patients with the Padua and IMPROVE Bleeding scores

SUMMARY:
FADOI (Italian Scientific Society of Hospital Internal Medicine) has planned to promote a multicenter cluster-randomized controlled clinical study in order to evaluate the effects of a systematic assessment of patients by using the Padua prediction score and the IMPROVE Bleeding score vs clinical judgement on the use of antithrombotic prophylaxis and clinical outcomes (thromboembolic and hemorrhagic events).

DETAILED DESCRIPTION:
The most recent guidelines suggest the use of prophylaxis in patients with a high thromboembolic risk, while taking into account the risk of bleeding.

It is known that patients admitted for acute pathology have an eight-fold higher incidence of thromboembolic events than the general population.

The Padua Prediction Score (PPS) is currently considered the best score available for the evaluation of thromboembolic risk in hospitalized patients, while the IMPROVE score was developed and validated for the assessment of bleeding risk in the same population of hospitalized patients.

In a recent study, data from the real world showed us how many of the patients admitted in Internal Medicine were at high thrombotic risk according to PPS and almost 90% of these were simultaneously at low hemorrhagic risk according to the IMPROVE score: in these patients pharmacological prophylaxis could therefore be prescribed during a safe stay.

Until now only a small prospective monocentric quasi-randomized study has shown that the use of systematic PPS reduces the incidence of thromboembolic events (symptomatic and non-symptomatic) upon discharge, compared to clinical judgment alone.

For these reasons, FADOI Foundation has promoted a multicenter controlled randomized cluster study in a real-life context among patients admitted to medical area departments. The aim of the study will be to analyze the effects of a systematic evaluation of patients (in centers that do not require the use of any score for the evaluation of thromboembolic risk), using the Padua Prediction Score (PPS) and the IMPROVE Bleeding score vs only clinical judgment for the use of antithrombotic prophylaxis and clinical outcomes (thromboembolic and haemorrhagic events). The main objective of the study is therefore to evaluate the effectiveness of a systematic evaluation of the thromboembolic and hemorrhagic risk in reducing the number of major complications in patients admitted to Internal Medicine, at a 90-day follow-up after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Hospitalized for any cause in Internal Medicine
3. Signature of informed consent

Exclusion Criteria:

1. Expected hospital stay < 48 h
2. Any indication for anticoagulant therapy
3. Life expectancy < 90 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2878 (Actual)
Dates: Start 2019-03-20 (Actual); Primary Completion 2021-05-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
The percentage of patients with major complications at a 90-day follow-up | 3 month from the discharge
  The percentage of patients with major complications (death, venous thromboembolism, major bleeding) at a 90-day follow-up in the group of patients who will be evaluated by means of the Padua and IMPROVE Bleeding scores vs those evaluated according to clinical judgment only

SECONDARY OUTCOMES:
Clinical outcomes at hospital discharge | Time of hospitalization until discharge, up to 5 weeks
  The percentage of patients with major complications (death, venous thromboembolism, major bleeding) at hospital discharge in the group of patients who will be evaluated by means of the Padua and IMPROVE Bleeding scores vs those evaluated according to clinical judgment only
Number of patients with antithrombotic prophylaxis during hospital stay and at discharge. | Time of hospitalization until discharge, up to 5 weeks
  All the clinical characteristics of the patient collected, are compared between the experimental group and the clinical judgment group to understand the choice of an antithrombotic prophylaxis

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Campanini, Study Director — Fadoi Foundation
Locations (35):
- Italy (35):
  - Ospedale di Casale Monferrato, Casale Monferrato, Alessandria
  - Ospedale "SS Antonio e Margherita", Tortona, Alessandria
  - Ospedale di Senigallia, Senigallia, Ancona
  - Ospedale di Molfetta, Molfetta, Bari
  - Ospedale Civile, Marcianise, Caserta
  - Ospedale di Ceva, Ceva, Cuneo
  - Ospedale di Mondovì, Mondovì, Cuneo
  - Osp. Casa Sollievo Della Sofferenza, San Giovanni Rotondo, Foggia
  - Ospedale Civile, Legnano, Milano
  - Ospedale di Magenta, Magenta, Milano
  - Ospedale Media Valle del Tevere, Todi, Perugia
  - Ospedale Generale di Zona, Lagonegro, Potenza
  - Ospedale San Marco, Grottaglie, Taranto
  - Ospedale di Rivoli, Rivoli, Torino
  - Ospedale San Giacomo Apostolo, Castelfranco Veneto, Treviso
  - Ospedale di Conegliano Veneto, Conegliano, Treviso
  - Ospedale "Luini Confalonieri", Luino, Varese
  - Ospedale di Borgosesia, Borgosesia, Vercelli
  - Ospedale Cardinal Massaia, Asti
  - Ospedale "Beato Angelo", Cosenza
  - Ospedale di Cremona, Cremona
  - Ospedale Santa Croce di Fano, Fano
  - E.O. Ospedali Galliera, Genova
  - Ospedale Maggiore Niguarda, Milan
  - Azienda Ospedaliera "Cardarelli", Napoli
  - Ospedale Fatebenefratelli, Napoli
  - Ospedale Silvestrini di Perugia, Perugia
  - Ospedale "Bianchi-Melacrino-Morelli", Reggio Calabria
  - Ospedale "S. Giovanni Addolorata", Roma
  - Ospedale "Vannini", Roma
  - Ospedale "San Paolo", Savona
  - Ospedale di Treviso, Treviso
  - Ospedale di Circolo "Macchi", Varese
  - Ospedale Sant'Andrea, Vercelli
  - Ospedale "S. Bortolo", Vicenza

REFERENCES:
- [Derived] Dentali F, Campanini M, Bonaventura A, Fontanella L, Zuretti F, Tavecchia L, Mumoli N, Gnerre P, Ventrella F, Giustozzi M, Valerio A, Fontanella A. The Use of Risk Scores for Thromboprophylaxis in Medically Ill Patients-Rationale and Design of the RICO trial. TH Open. 2024 Jan 12;8(1):e55-e60. doi: 10.1055/a-2209-4708. eCollection 2024 Jan. PMID 38222040